CLINICAL TRIAL: NCT06023771
Title: Drainage and Debridement of Local Complications of Acute Pancreatitis: A Single-center Real-world Prospective Study
Brief Title: Invasive Intervention of Local Complications of Acute Pancreatitis
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K4433
Record Dates: First submitted 2023-08-17; First posted 2023-09-05 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute pancreatitis requiring invasive intervention: Single-center cohort of acute pancreatitis patients requiring invasive intervention for the treatment of local complications during the whole course of disease.
  Interventions: Procedure: Invasive intervention for acute pancreatitis

INTERVENTIONS:
Procedure: Invasive intervention for acute pancreatitis — Invasive interventions include drainage (endoscopic transmural drainage, imaging-guided percutaneous catheter drainage) and debridement (endoscopic debridement, videoscopic assisted retroperitoneal debridement, laparoscopic surgical debridement, open surgical debridement).

SUMMARY:
Strategies for invasive intervention in acute pancreatitis include sequential or combined use of multiple drainage and debridement modalities. The more widely used is the step-up approach, which requires an individualized and multidisciplinary (internal medicine, interventional radiology, endoscopy, surgery, critical care medicine, and nutritionists) approach. The available evidence from randomized controlled studies is from highly selected subject populations, and it is unclear whether the results can be applied to complex clinical situations in real clinics, and the optimal strategy for drainage of peripancreatic lesions in different patients still needs to be evaluated in the real world. This study intends to establish a prospective single-center cohort for real-world analysis to collect comprehensive clinic information and clinical outcomes, to evaluate the effectiveness and safety of existing intervention strategies, especially the timing and modality of interventions, in real-world clinical practice, and to explore the key factors affecting patient prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Admission diagnosis of acute pancreatitis;
* Localized complications confirmed by imaging examinations;
* Voluntary participation in the study and signing of an informed consent form.

Exclusion Criteria:

* Improved with conservative treatment without invasive interventions for local complications during hospitalization.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized acute pancreatitis patients requiring invasive interventions.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Major complications or death | Day 1 from admission until 6 months after discharge
  A composite of major complications (i.e., new-onset multiple organ failure or systemic complications, enterocutaneous fistula or perforation of a visceral organ requiring intervention, or intraabdominal bleeding requiring intervention) or death during admission or during the 6 months after discharge.

SECONDARY OUTCOMES:
Organ failure | Day 1 from admission until 6 months after discharge
  New-onset ( not present at any time in the 24 hours before first intervention) pulmonary failure, circulatory failure, or renal failure
Systemic complication | Day 1 from admission until 6 months after discharge
  New-onset ( not present at any time in the 24 hours before first intervention) systematic complications such as disseminated intravascular coagulation, severe metabolic disturbance, and gastrointestinal bleeding
Enterocutaneous fistula | Day 1 from admission until 6 months after discharge
  Secretion of fecal material from a percutaneous drain or drainage canal after removal of drains or from a surgical wound, either from small or large bowel; confirmed by imaging or during surgery
Perforation of visceral organ | Day 1 from admission until 6 months after discharge
  Perforation requiring surgical, radiologic, or endoscopic intervention
Intraabdominal bleeding | Day 1 from admission until 6 months after discharge
  Requiring surgical, radiologic, or endoscopic intervention
Pancreatic fistula | Day 1 from admission until 6 months after discharge
  Output, through a percutaneous drain or drainage canal after removal of drains or from a surgical wound, of any measurable volume of fluid with an amylase content >3 times the serum amylase level
New-onset diabetes | Day 1 from admission until 6 months after discharge
  Insulin or oral antidiabetic drugs required 6 mo after discharge; this requirement was not present before onset of pancreatitis
Use of pancreatic enzymes | Day 1 from admission until 6 months after discharge
  Oral pancreatic-enzyme supplementation required to treat clinical symptoms of steatorrhea 6 mo after discharge; this requirement was not present before onset of pancreatitis
Length of hospitalization | Day 1 from admission until the 1 day of discharge
  Total days of hospitalization for the management of acute pancreatitis
Length of intesive care | Day 1 from admission until the 1 day of discharge
  Total days in intesive care unit for the management of acute pancreatitis
Total direct medical costs and indirect costs | Day 1 from admission until the 1 day of discharge
  Total direct medical costs and indirect costs during admission

CONTACTS AND LOCATIONS:
Overall Officials: Dong Wu, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No